CLINICAL TRIAL: NCT04493320
Title: 1/2-Dopaminergic Dysfunction in Late-Life Depression (The D3 Study)
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Study terminated by sponsor (NIMH)
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); Vanderbilt University Medical Center (Other); Columbia University (Other); Emory University (Other)
Responsible Party: Principal Investigator, Bret Rutherford, Associate Professor of Clinical Psychiatry, New York State Psychiatric Institute
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 7976; R01MH123660-01 (NIH)
Record Dates: First submitted 2020-07-27; First posted 2020-07-30 (Actual); Results first posted 2023-05-22 (Actual); Last update posted 2023-05-22 (Actual); Status verified 2023-05

CONDITIONS: Depression; Cognitive Impairment; Gait Impairment
MeSH Terms: conditions — Depression; Cognitive Dysfunction | interventions — carbidopa, levodopa drug combination; Levodopa

STUDY DESIGN:
Intervention Model Description: Double blind crossover study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- L-DOPA, Then Placebo (Experimental): Step 1 (3 Weeks): Participants will first receive 150 mg of L-DOPA daily in Week 1, 300 mg of L-DOPA in Week 2, and 450 mg L-DOPA in Week 3.
  Participants will then enter a 1 week taper period.
  Step 2 (3 Weeks): Participants will receive L-DOPA matching placebo tablets daily.
  Participants will then enter a 1-week taper period.
  Interventions: Drug: Carbidopa/levodopa; Drug: Placebo
- Placebo, Then L-DOPA (Experimental): Step 1 (3 Weeks): Participants will receive 3 L-DOPA matching placebo tablets daily. Participants will then enter a 1-week taper period.
  Step 2 (3 Weeks): Participants will first receive 150 mg of L-DOPA daily in Week 1, 300 mg of L-DOPA in Week 2, and 450 mg L-DOPA in Week 3.
  Participants will then enter a 1-week taper period.
  Interventions: Drug: Carbidopa/levodopa; Drug: Placebo

INTERVENTIONS:
Drug: Carbidopa/levodopa — 150-450mg carbidopa/levodopa 3 times daily
  Other Names: L-DOPA; Sinemet
Drug: Placebo — Carbidopa/levodopa-matched placebo tablet 3 times daily
  Other Names: Placebo tablet

SUMMARY:
Growing evidence suggests that dopamine contributes to key cognitive, emotional, and motor functions across the lifespan. In Late-Life Depression (LLD), dysfunction in these areas is common, predicts poor outcomes, and manifests as difficulties in motivation and effort along with cognitive and gait impairment. While studies of dopamine function in early and midlife depression primarily focus on individuals' ability to feel pleasure and respond to rewards, they often exclude the cognitive and physical function domains relevant for older adults despite a recognized decline in dopamine function with normal aging. The objectives of this collaborative R01 proposal between Columbia University/New York State Psychiatric Institute and Vanderbilt University Medical Center are to: 1) characterize dopaminergic dysfunction in LLD across cognitive, emotional, and motor domains at several levels of analysis (cellular Positron Emission Tomography [PET], circuit Magnetic Resonance Imaging [MRI], and behavioral / self-report); and 2) examine the responsivity of dopamine-related circuits and behavior to stimulation with carbidopa/levodopa (L-DOPA).

DETAILED DESCRIPTION:
Supported by pilot data, this project builds on past work demonstrating that dopamine function declines with aging, that dopaminergic dysfunction contributes to deficits in behavior, and that L-DOPA administration improves cognitive and motor performance. The long-term goal of this line of research is to determine how dopaminergic dysfunction contributes to clinical presentations of LLD, how responsive behavioral symptoms are to modulation of dopamine function, and to identify novel targets for future interventions. Investigator's approach is to enroll 30 psychiatrically healthy elders and 60 depressed elders at Columbia/NYSPI exhibiting either slowed processing speed or slowed gait speed. Participants will undergo thorough clinical evaluations and complete PET imaging measuring different aspects of the brain's dopamine system, neuromelanin-sensitive MRI measurement of longterm dopamine transmission, functional MRI focused on effort-based decision making and reward processing, a comprehensive neurocognitive evaluation, a physical performance evaluation, and measurement of inflammatory markers. To assess responsivity of the dopamine system to modulation, depressed subjects then will be randomized to L-DOPA or placebo for 3 weeks, followed by repeat multimodal MRI and cognitive/behavioral assessments. In a second phase, participants will receive the opposite intervention for an additional 3 weeks followed by clinical and cognitive assessments only. This proposal is significant and innovative, as no prior published study has comprehensively examined dopamine-dependent behaviors in LLD. This will inform treatment approaches focusing on facilitating cognition and movement, reducing the effort cost of voluntary behavior, and promoting behavioral activation.

ELIGIBILITY:
Inclusion Criteria:

Depressed Subjects:

1. Age 60 years or older (female subjects will be post-menopausal by virtue of their age, but last menstrual period month and year will be documented in the study database)
2. Diagnosis and Statistical Manual (DSM-5) diagnosis of Major Depressive Disorder (MDD) or Persistent Depressive Disorder (PDD)
3. Montgomery Asberg Depression Rating Scale Score (MADRS) >=15
4. Decreased processing speed or decreased gait speed
5. Capable of providing informed consent and complying with study procedures
6. Alternative standard treatments for MDD or PDD have been discussed and the individual agrees to be involved in an experimental treatment

Psychiatrically Healthy Elders:

1. Age 60 years or older years old
2. MADRS < 8
3. Capable of providing informed consent and complying with study procedures

Exclusion Criteria:

Depressed Subjects:

1. Diagnosis of Substance Use Disorder (excluding Tobacco Use Disorder) in the past 12 months
2. History of psychosis (except brief psychosis associated with transient medical conditions [e.g., delirium, urinary tract infection, etc], psychotic disorder, mania, or bipolar disorder.
3. Primary neurological disorder, including dementia, stroke, Parkinson's disease, or epilepsy.
4. Mini Mental State Examination (MMSE) < 24
5. MADRS suicide item >4 or other indication of acute suicidality
6. Current or recent (within the past 2 weeks) treatment with antidepressants, antipsychotics, or mood stabilizers
7. History of hypersensitivity, allergy, or intolerance to L-DOPA
8. Any physical or intellectual disability adversely affecting ability to complete assessments.
9. Acute, severe, or unstable medical illness
10. Mobility limiting osteoarthritis of any lower extremity joints, symptomatic lumbar spine disease, or history of joint replacement or spine surgery that limits mobility
11. Contraindication to MRI scanning (Metal implants, pacemaker, metal prostheses, metal orthodontic appliances in the body unless there is confirmation that the substance is MRI compatible.)
12. History of significant radioactivity exposure (nuclear medicine studies or occupational exposure)
13. Has a medical condition managed with medication and/or device and the managing physician considers the condition and/or its management a contraindication to the research use of L-DOPA in this participant

Psychiatrically Healthy Elders:

1. Any personal history of DSM-5 disorder
2. Family history of MDD in first-degree relative
3. Plus, Exclusion criteria 8-12 above

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2021-02-10 (Actual); Primary Completion 2021-10-27 (Actual); Study Completion 2021-10-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bret R Rutherford, MD, Principal Investigator — New York State Psychiatric Institute
Locations (1):
- New York State Psychiatric Institute, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: In total, 5 depressed subjects were enrolled. Of the 5 enrolled, 1 subject was found to be ineligible. Thus, 5 participants enrolled and 4 were assigned to a treatment group and began the study.
Groups:
- L-DOPA, Then Placebo: Step 1 (3 Weeks): Participants will first receive 150 mg of L-DOPA daily in Week 1, 300 mg of L-DOPA in Week 2, and 450 mg L-DOPA in Week 3.
  Participants will then enter a 1 week taper period.
  Step 2 (3 Weeks): Participants will receive L-DOPA matching placebo tablets daily.
  Participants will then enter a 1-week taper period.
  Carbidopa/levodopa: 150-450mg carbidopa/levodopa 3 times daily
  Placebo: Carbidopa/levodopa-matched placebo tablet 3 times daily
- Placebo, Then L-DOPA: Step 1 (3 Weeks): Participants will receive 3 L-DOPA matching placebo tablets daily. Participants will then enter a 1-week taper period.
  Step 2 (3 Weeks): Participants will first receive 150 mg of L-DOPA daily in Week 1, 300 mg of L-DOPA in Week 2, and 450 mg L-DOPA in Week 3.
  Participants will then enter a 1-week taper period.
  Carbidopa/levodopa: 150-450mg carbidopa/levodopa 3 times daily
  Placebo: Carbidopa/levodopa-matched placebo tablet 3 times daily
Period: Overall Study
Arm/Group | L-DOPA, Then Placebo | Placebo, Then L-DOPA
Started | 2 | 2
Completed | 1 | 1
Not Completed | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | L-DOPA, Then Placebo | Placebo, Then L-DOPA | Total
Number analyzed (Participants) | 2 | 2 | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 74.5 (16.3) | 65.5 (7.8) | 70.0 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1
  Male | 2 | 1 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 2 | 2 | 4
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 2 | 2 | 4
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Montgomery Asberg Depression Rating Scale [Mean (Standard Deviation); unit: units on a scale] | 24.5 (5.0) | 36.5 (12.0) | 25.5 (7.6)
Clinical Global Impressions--Severity [Mean (Standard Deviation); unit: units on a scale] — The Clinical Global Impressions--Severity (CGI-S) scale measures the clinician's assessment of global illness severity. Scores range from 1 (normal, not at all ill) to 7 (among the most extremely ill patients). Higher scores denote more severe illness.
  units on a scale | 5.0 (0.0) | 4.0 (0.0) | 4.3 (0.6)
Quick Inventory for Depressive Symptomatology [Mean (Standard Deviation); unit: units on a scale] | 10.0 (0.0) | 15.0 (4.2) | 13.3 (4.2)

OUTCOME MEASURES:

1. Primary Outcome: Change in Effort Expenditure for Rewards Task (EEfRT) Following Step 1
Description: In this task participants decide whether to work harder for a larger reward (high number of finger presses with their pinky) or expend less energy (low number of presses with a dominant index finger) for a lesser reward, with lower rewards being $1 dollar and higher rewards ranging from $1.20 to $5. Participants receive information about the probability of winning on each trial regardless of their pick and one trial from each run is randomly picked for payout. The primary output on this task is the percentage of time participants choose the high cost / high reward option on the EEfRT. Because the full sample was not enrolled and the results are considered unreliable, no statistical analysis was performed other than calculating means and standard deviations.
  This task was not completed following Step 2 of the study, so there are no EEfRT data reported for change in task performance following Step 2.
Time Frame: Change from Baseline to 3 weeks (post Step 1)
Population: Participants with Baseline and Week 3 data available were analyzed
Measure: Mean (Standard Deviation); unit: percentage of high effort choices
Arm/Group | L-DOPA, Then Placebo | Placebo, Then L-DOPA
Number analyzed (Participants) | 1 | 2
percentage of high effort choices | 0.18 (NA) — Standard Deviation is not calculable for 1 participant. | 0.0 (0.0)

2. Primary Outcome: Change in Digit Symbol Test Following Step 1
Description: The Digit Symbol test is a neuropsychological test measuring information processing speed. It consists of digit-symbol pairs (e.g. 1/-,2/┴ ... 7/Λ,8/X,9/=) followed by a list of digits. Under each digit the subject should write down the corresponding symbol as fast as possible. The number of correct symbols within the allowed time is measured. Score ranges from 0-133, with higher scores indicating higher information processing speed. Because the full sample was not enrolled and the results are considered unreliable, no statistical analysis was performed other than calculating means and standard deviations.
Time Frame: Change from Baseline to 3 weeks (post Step 1)
Population: Participants with Baseline and Week 3 data available were analyzed
Measure: Mean (Standard Deviation); unit: Number of items correctly completed
Arm/Group | L-DOPA, Then Placebo | Placebo, Then L-DOPA
Number analyzed (Participants) | 2 | 2
Number of items correctly completed | -0.5 (2.1) | 9.0 (7.1)

3. Primary Outcome: Change in Digit Symbol Test Following Step 2
Description: as for outcome 2
Time Frame: Change from Week 3 to Week 7 (post-Step 2)
Population: Participants with Week 3 and Week 7 data available were analyzed
Measure: Number; unit: Number of items correctly completed
Arm/Group | L-DOPA, Then Placebo | Placebo, Then L-DOPA
Number analyzed (Participants) | 1 | 1
Number of items correctly completed | 5.0 | 4.0

4. Primary Outcome: Change in Pattern Comparison Test Following Step 1
Description: This test required participants to identify whether two visual patterns are the "same" or "not the same" (responses were made by pressing a "yes" or "no" button). Patterns were either identical or varied on one of three dimensions: color (all ages), adding/taking something away (all ages), or one versus many. Scores reflect the number of correct items completed in 90 s, with scores ranging from a minimum of 0 to a maximum of 30. Items were designed to minimize the number of errors that were made. Because the full sample was not enrolled and the results are considered unreliable, no statistical analysis was performed other than calculating means and standard deviations.
Time Frame: Change from Baseline to 3 weeks (post Step 1)
Population: Participants with Baseline and Week 3 data available were analyzed
Measure: Mean (Standard Deviation); unit: Number of items correctly completed
Arm/Group | L-DOPA, Then Placebo | Placebo, Then L-DOPA
Number analyzed (Participants) | 2 | 2
Number of items correctly completed | -1.0 (1.4) | 1.75 (1.1)

5. Primary Outcome: Change in Pattern Comparison Test Following Step 2
Description: as for outcome 4
Time Frame: Change from Week 3 to Week 7 (post-Step 2)
Population: Participants with Week 3 and Week 7 data available were analyzed
Measure: Number; unit: Number of items correctly completed
Arm/Group | L-DOPA, Then Placebo | Placebo, Then L-DOPA
Number analyzed (Participants) | 1 | 1
Number of items correctly completed | 1.0 | -3.5

6. Primary Outcome: Change in Letter Comparison Test Following Step 1
Description: Subjects were asked to determine whether two strings of letters are the same or different. There are 3 pages and the subject is given 30 seconds per page. Scoring is based on the number answered correctly. Scores range from 0 to 21, with the higher the number, the better the score. Because the full sample was not enrolled and the results are considered unreliable, no statistical analysis was performed other than calculating means and standard deviations.
Time Frame: Change from Baseline to 3 weeks (post Step 1)
Population: Participants with Baseline and Week 3 data available were analyzed
Measure: Mean (Standard Deviation); unit: Number of items correctly completed
Arm/Group | L-DOPA, Then Placebo | Placebo, Then L-DOPA
Number analyzed (Participants) | 2 | 2
Number of items correctly completed | -0.5 (0.0) | -0.25 (2.5)

7. Primary Outcome: Change in Letter Comparison Test Following Step 2
Description: as for outcome 6
Time Frame: Change from Week 3 to Week 7 (post-Step 2)
Population: Participants with Week 3 and Week 7 data available were analyzed
Measure: Number; unit: Number of items correctly completed
Arm/Group | L-DOPA, Then Placebo | Placebo, Then L-DOPA
Number analyzed (Participants) | 1 | 1
Number of items correctly completed | 0.5 | -1.5

8. Primary Outcome: Change in Single Task Gait Speed Test Following Step 1
Description: Patients' gait was assessed as walking speed in cm/s on a 15' walking course. Patients walked at their usual or normal speed for a total of 27' (starting and ending at a point 6 feet prior to and after the 15' course to eliminate acceleration and deceleration effects). Two trials were completed, and gait speed was based on the average of 2 trials. Because the full sample was not enrolled and the results are considered unreliable, no statistical analysis was performed other than calculating means and standard deviations.
Time Frame: Change from Baseline to 3 weeks (post Step 1)
Population: Participants with Baseline and Week 3 data available were analyzed
Measure: Mean (Standard Deviation); unit: cm/s
Arm/Group | L-DOPA, Then Placebo | Placebo, Then L-DOPA
Number analyzed (Participants) | 2 | 2
cm/s | 4.6 (5.9) | 11.9 (11.2)

9. Primary Outcome: Change in Single Task Gait Speed Test Following Step 2
Description: as for outcome 8
Time Frame: Change from Week 3 to Week 7 (post-Step 2)
Population: Participants with Week 3 and Week 7 data available were analyzed
Measure: Number; unit: cm/s
Arm/Group | L-DOPA, Then Placebo | Placebo, Then L-DOPA
Number analyzed (Participants) | 1 | 1
cm/s | -17.2 | 7.0

10. Primary Outcome: [18F]-FDOPA PET Measure in Striatal Region of Interest
Description: [18F]-FDOPA PET quantifies dopamine synthesis capacity in specific brain regions. Lower [18F]-FDOPA uptake in the striatum has been associated with increased depression severity and worse cognitive and motor function in patients. Because [18F]-FDOPA uptake may be sensitive to deficits in dopamine synthesis capacity in older depressed patients, in this study depressed participants at baseline underwent a PET scan to quantify relative [18F]-FDOPA influx rate in the nucleus accumbens bilaterally. Time activity curves (TACs) were extracted within the nucleus accumbens region of interest (ROI) as the average radioactivity in the ROI over time. The occipital lobe, which has the lowest dopamine concentration in the brain, was used as the "reference region" to yield the Kocc measure of [18F]-FDOPA influx rate. Higher [18F]-FDOPA influx rate (kocc) numbers indicate greater relative influx rate and therefore greater dopamine synthesis capacity.
Time Frame: Baseline (prior to LDOPA or placebo administration)
Population: Participants who had a baseline [18F]-FDOPA PET scan
Measure: Number; unit: min^-1
Arm/Group | L-DOPA, Then Placebo | Placebo, Then L-DOPA
Number analyzed (Participants) | 1 | 0
min^-1 | 0.0107 |

11. Secondary Outcome: Change in Montgomery Asberg Depression Rating Scale Following Step 1
Description: Secondary outcome measured by the total score of the clinician rated MADRS, a measure of depression severity. The MADRS total score range is 0-60, where higher scores indicate greater depression severity. Because the full sample was not enrolled and the results are considered unreliable, no statistical analysis was performed other than calculating means and standard deviations.
Time Frame: Change from Baseline to 3 weeks (post Step 1)
Population: Participants with Baseline and Week 3 data available were analyzed
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | L-DOPA, Then Placebo | Placebo, Then L-DOPA
Number analyzed (Participants) | 2 | 2
units on a scale | -1.0 (9.9) | -3.0 (2.8)

12. Secondary Outcome: Change in Montgomery Asberg Depression Rating Scale Following Step 2
Description: Secondary outcome measured by the total score of the clinician rated MADRS, a measure of depression severity. The MADRS total score range is 0-60, where higher scores indicate greater depression severity. In contrast to other measures, which were not available at Week 4, Week 4 was selected as the baseline for post-Step 2 change on the MADRS since it followed the taper period taking place between study Steps. Because the full sample was not enrolled and the results are considered unreliable, no statistical analysis was performed other than calculating means and standard deviations.
Time Frame: Change from Week 4 to Week 7 (post-Step 2)
Population: Participants with Week 4 and Week 7 data available were analyzed
Measure: Number; unit: units on a scale
Arm/Group | L-DOPA, Then Placebo | Placebo, Then L-DOPA
Number analyzed (Participants) | 1 | 1
units on a scale | 4.0 | 2.0

13. Secondary Outcome: Change in Quick Inventory for Depressive Symptomatology (QIDS) Following Step 1
Description: QIDS-16-item, a participant-rated measure of depressive symptomatology. The total score ranges from 0 to 27, with higher scores indicative of greater severity. Because the full sample was not enrolled and the results are considered unreliable, no statistical analysis was performed other than calculating means and standard deviations.
Time Frame: Change from Baseline to 3 weeks (post Step 1)
Population: Participants with Baseline and Week 3 data available were analyzed
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | L-DOPA, Then Placebo | Placebo, Then L-DOPA
Number analyzed (Participants) | 1 | 2
units on a scale | -1.0 (0.0) | -5.0 (5.7)

14. Secondary Outcome: Change in Quick Inventory for Depressive Symptomatology (QIDS) Following Step 2
Description: QIDS-16-item, a participant-rated measure of depressive symptomatology. The total score ranges from 0 to 27, with higher scores indicative of greater severity. In contrast to other measures, which were not available at Week 4, Week 4 was selected as the baseline for post-Step 2 change on the QIDS since it followed the taper period taking place between study Steps. Because the full sample was not enrolled and the results are considered unreliable, no statistical analysis was performed other than calculating means and standard deviations.
Time Frame: Change from Week 4 to Week 7 (post-Step 2)
Measure: Number; unit: units on a scale
Arm/Group | L-DOPA, Then Placebo | Placebo, Then L-DOPA
Number analyzed (Participants) | 1 | 1
units on a scale | -1.0 | 0.0

ADVERSE EVENTS:
Time Frame: Subjects were monitored over a period of 7 weeks.
Groups:
- L-DOPA: This trial entailed the administration of either L-DOPA or placebo in Step 1, followed by crossover to the other treatment assignment in Step 2 (i.e., L-DOPA followed by placebo or placebo followed by L-DOPA). Adverse events are grouped here by treatment assignment (L-DOPA or placebo). This arm pertains to the administration of L-DOPA in Step 1 and Step 2 of the study.
- Placebo: This trial entailed the administration of either L-DOPA or placebo in Step 1, followed by crossover to the other treatment assignment in Step 2 (i.e., L-DOPA followed by placebo or placebo followed by L-DOPA). Adverse events are grouped here by treatment assignment (L-DOPA or placebo). This arm pertains to the administration of placebo in Step 1 and Step 2 of the study.
Arm/Group | L-DOPA | Placebo
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/3
Other Adverse Events (participants affected / at risk) | 3/4 | 2/3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | L-DOPA (N=4) | Placebo (N=3)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 1 (2)
Dizziness (Vascular disorders) | 1 (1) | 1 (1)
Increased blood pressure (Vascular disorders) | 1 (1) | 0 (0)
Faintness (General disorders) | 0 (0) | 1 (1)
Drowsiness (Psychiatric disorders) | 0 (0) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Data collected in the trial have been presented as required but are considered unreliable.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2020-07-24): https://cdn.clinicaltrials.gov/large-docs/20/NCT04493320/Prot_000.pdf
  • Statistical Analysis Plan (2019-10-03): https://cdn.clinicaltrials.gov/large-docs/20/NCT04493320/SAP_001.pdf
  • Informed Consent Form (2020-07-24): https://cdn.clinicaltrials.gov/large-docs/20/NCT04493320/ICF_002.pdf